CLINICAL TRIAL: NCT05879978
Title: A Phase I, Non-randomized, Open-label, Multi-center Dose Escalation Trial of Obrixtamig (BI 764532) Combined With Ezabenlimab in Patients With Small Cell Lung Carcinoma and Other Neuroendocrine Neoplasms Expressing DLL3
Brief Title: A Study to Test How Well Different Doses of Obrixtamig (BI 764532) in Combination With Ezabenlimab Are Tolerated by People With Small Cell Lung Cancer and Other Neuroendocrine Tumours That Are Positive for DLL3
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1438-0002; 2022-502728-30-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-05-25; First posted 2023-05-30 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Small Cell Lung Carcinoma (SCLC); Neuroendocrine Neoplasms
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- obrixtamig + ezabenlimab treatment group (Experimental): Successive cohorts of patients will receive increasing doses of obrixtamig in combination with ezabenlimab until the maximum tolerated dose (MTD) is reached, or upon decision of Dose Escalation Committee (DEC).
  Interventions: Drug: Obrixtamig; Drug: Ezabenlimab

INTERVENTIONS:
Drug: Obrixtamig — Obrixtamig
  Other Names: BI 764532
Drug: Ezabenlimab — Ezabenlimab

SUMMARY:
This study is open to adults with small cell lung cancer and other neuroendocrine tumours that are positive for the tumour marker Delta-like 3 (DLL3). The study is in people with advanced cancer for whom previous treatment was not successful or no standard treatment exists.

The purpose of this study is to find out the highest dose of obrixtamig that people can tolerate when taken together with another medicine called ezabenlimab. Obrixtamig and ezabenlimab may help the immune system fight cancer. Participants get obrixtamig and ezabenlimab as infusions into a vein.

If there is benefit for the participants and if they can tolerate it, the treatment is given for a maximum of 3 years. During this time, participants visit the study site about every week. The visits also depend on the response to the treatment. At the study visits, the doctors check the health of the participants, take necessary laboratory tests, and note any health problems that could have been caused by the study treatment.

ELIGIBILITY:
Inclusion criteria

1. Age ≥18 years
2. Signed and dated, written informed consent form (main ICF) in accordance with ICH-GCP and local legislation prior to any trial-specific procedures, sampling, or analyses.
3. Diagnosed with locally advanced, metastatic or relapsed cancer not amenable to curative treatment of the following histologies:

   * Small cell lung carcinoma (SCLC)
   * Large cells neuroendocrine lung carcinoma(LCNEC)
   * Neuroendocrine carcinoma (NEC) or small cell carcinoma of any other origin

     * Tumours must be positive for Delta-like 3 (DLL3) expression (on archived tissue) according to central pathology review in order to start obrixtamig.
     * Patients with tumors with mixed histologies for any above type are eligible only if neuroendocrine carcinoma/small tumor cells component is predominant and represent at least 50% of the overall tumor tissue.
4. Patient who failed conventional treatment or for whom no therapy of proven efficacy exists or who is not eligible for established treatment options. Patient must have exhausted available treatment options known to prolong survival for their disease. Previous therapies should include at least one line of platinum-based chemotherapy.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. At least one evaluable lesion outside of Central Nervous System (CNS) as defined per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
7. Subjects with brain metastases are eligible provided they meet the following criteria:

   * radiotherapy or surgery for brain metastases was completed at least 2 weeks or 4 weeks respectively, prior to the first administration of obrixtamig
   * patient is off steroids for at least 7 days (physiologic doses of steroids are permitted), and the patient is off anti-epileptic drugs for at least 7 days or on stable doses of anti-epileptic drugs for malignant CNS disease.
8. Male or female patients. Women of childbearing potential (WOCBP)1 and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.These methods must be used during the study and for at least 3 months after the last dose of obrixtamig. A list of contraception methods meeting these criteria is provided in the patient information.

Further inclusion criteria apply.

Exclusion criteria

1. Previous treatment with T-cell-engager (TcE) or cell therapies targeting DLL3. Other DLL3 targeting agents (like RovaT) are allowed only if DLL3 positivity is documented after completion of treatment with DLL3 targeting agent in post-treatment biopsy.
2. Previous or concomitant malignancies other than the one treated in this trial within the last 2 years except:

   * effectively treated non-melanoma skin cancers
   * effectively treated carcinoma in situ of the cervix
   * effectively treated ductal carcinoma in situ
   * other effectively treated malignancy that is considered cured by local treatment
3. Major injuries and/or surgery or bone fracture within 28 days of first dose obrixtamig, or planned surgical procedures
4. Known leptomeningeal disease or spinal cord compression due to metastatic disease
5. Anticoagulant treatment that cannot be safely interrupted based on opinion of the investigator if medically needed
6. Patients who have been febrile, have had leukocytosis, or any clinical signs of infection within 48 h prior to randomization/start of trial treatment are not eligible. Oral or intravenous antimicrobials for management of fungal, bacterial, viral, or other infection are prohibited within 7 days prior to randomization/start of trial treatment. The use of antimicrobials for routine infection prophylaxis is acceptable
7. Severe acute respiratory syndrome coronavirus 2 (SARS COV2) infection within 2 weeks prior to study entry (confirmed via Polymerase chain reaction (PCR) test or other applicable test as per local requirements) or suspected SARS-CoV-2 infection as per physician assessment, or close contact (within 1 week) with an individual with confirmed SARS-CoV-2 infection
8. Any of the following known laboratory evidence of hepatitis virus infection:

   * Positive results of hepatitis B surface (HBs) antigen
   * Presence of hepatitis B core (HBc) antibody together with hepatitis B virus (HBV)-Deoxyribonucleic Acid (DNA)
   * Presence of hepatitis C Ribonucleic acid (RNA) Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicities (DLTs) in the Maximum Tolerated Dose (MTD) evaluation period | up to 19 months

SECONDARY OUTCOMES:
Occurrence of DLTs during the on-treatment period | up to 19 months
Objective response, defined as best overall response of complete response (CR) or partial response (PR) | up to 19 months
  Objective response, defined as best overall response of complete response (CR) or partial response (PR), where best overall response is determined by the investigator's assessment according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 in patients with measurable disease from date of first treatment administration until the earliest of disease progression, death or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow-up or withdrawal of consent
Cmax (maximum measured concentration of obrixtamig) | up to 19 months
Cmax (maximum measured concentration of ezabenlimab) | up to 19 months
AUCτ (area under the concentration-time curve of obrixtamig over a uniform dosing interval τ) | up to 19 months
AUCτ (area under the concentration-time curve of ezabenlimab) over a uniform dosing interval τ) | up to 19 months

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UNIV UZ Gent, Ghent
- France (3):
  - HOP Louis Pradel, Bron
  - CTR François Baclesse, Caen
  - INS Claudius Regaud IUCT-Oncopole, Toulouse
- Germany (2):
  - Technische Universität Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt
- National Cancer Center Hospital, Tokyo, Chuo-ku, Japan

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com